CLINICAL TRIAL: NCT00194012
Title: Aripiprazole in At-Risk Children With Symptoms of Bipolar Disorder
Brief Title: Study of Aripiprazole (Abilify) Versus Placebo in Children With Subsyndromal Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Robert L Findling, MD, Director, Division of Child and Adolescent Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: At Risk
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole-Randomized Phase (Active Comparator): Patients randomly assigned to aripiprazole received medication in pill form with dosing at 2mg, 5mg, 7mg, 10mg, 12mg or 15mg depending on their response.
  Interventions: Drug: Aripiprazole
- Placebo-Randomized Phase (Placebo Comparator): Patients randomly assigned to placebo received pills/dosing made to look identical to the aripiprazole.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Addressed in arm description.
  Other Names: Abilify
  Arms: Aripiprazole-Randomized Phase
Drug: Placebo — Addressed in arm description.
  Arms: Placebo-Randomized Phase

SUMMARY:
The purpose of this study is to test the effectiveness and tolerability/safety of aripiprazole (Abilify) in children with subsyndromal symptoms of bipolar disorder who also have a parent with bipolar disorder and other family member with a mood disorder.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled, parallel-arm, randomized clinical trial that will last up to 12 weeks.

This placebo-controlled portion will be followed by a 6-week open label extension/stabilization phase. In order to be eligible for participation in the extension/stabilization phase, subjects must: 1) in the investigator's opinion have had no dose-limiting side effects likely to be attributable to aripiprazole (APZ); 2) participated in the blinded portion of the clinical trial for a minimum of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ages 5-17 years (inclusive)
* Patients, who in the investigator's opinion have substantial symptoms of mania, depression, or both within the past 2 weeks such that treatment with a pharmacological agent is warranted
* Currently meets Diagnostic Statistical Manual of Mental Disorders (DSM-IV) criteria for either cyclothymia, or bipolar disorder not otherwise specified (BP NOS) based on the results of both a semi-structured diagnostic research assessment, Present and Lifetime Version (K-SADS-Present and Lifetime (PL) supplemented with sections from the Washington University K-SADS) (Geller et al., 2001; Kaufman et al., 1997) and a clinical interview with a child and adolescent psychiatrist.
* Offspring of a parent with a bipolar spectrum disorder (based on the results of either the Mini International Neuropsychiatric Interview (MINI)(Sheehan et al., 1998) or the Family History Method (FH-RDC)(Andreasen et al., 1977)
* Has another first or second degree relative with a mood disorder determined by the results of either the MINI or the FH-RDC
* Has participated in at least 4 sessions of psychotherapy specifically focused on the symptoms/management of pediatric mood disorder and continues to have clinically significant symptomatology

Exclusion Criteria:

* Patients who have a history of intolerance to APZ at doses of 0.1mg/kg/day
* Patients who have experienced a manic episode with documented treatment with APZ monotherapy at a dose of 0.2 mg/kg/day
* Patients with an active neurological/medical disorder for which treatment with APZ would be contraindicated
* Patients with clinical evidence of autistic disorder, Asperger's disorder, Rett's syndrome or other pervasive developmental disorder
* Patients with clinical evidence of mental retardation
* Patients who are known to be allergic or hypersensitive to aripiprazole
* Patients who are unable to swallow pills/capsules
* Patients for whom the need for hospitalization during the course of the study appears likely
* Patients who have started a new psychotherapeutic intervention within less than 4 weeks of randomization
* Patients who have a general medical or neurological condition (including clinically significant abnormalities on screening laboratories) that may be considered to be the etiology of the patient's mood disorder
* Patients who have a general medical or neurological condition for which treatment with an atypical antipsychotic would be contraindicated (e.g. tardive dyskinesia)
* Patients who have a general medical or neurological condition that could interfere with the interpretation of clinical response to APZ treatment
* Patients taking psychotropic agents (other than psychostimulants) within one week of baseline (2 weeks for fluoxetine; 3 days for psychostimulants)
* Patients with a suicide attempt requiring medical/psychiatric care within the past 6 months
* Has met DSM-IV criteria for drug/alcohol abuse or dependence within the past 6 months
* Females who are currently pregnant or lactating
* Sexually active females, who in the investigators' opinion are not using an adequate form of birth control

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2004-08; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Findling, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- University Hospitals Case Medical Center - Walker Building, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited beginning 8/2004 with follow up interviews completed 5/2012. Families were recruited from an outpatient child/adolescent psychiatric research center and an adult mood disorders program at University Hospitals, Case Medical Center.
Pre-assignment Details: After screening and baseline assessments study participants were assigned to aripiprazole or placebo. Treatment was initiated at a dose of 0.1mg/kg/d. The dose could be increased by approximately 0.05 mg/kg/d at each study visit if patient experienced residual symptomology with no intolerable side effect to maximum dose 15mg/d.
Groups:
- Aripiprazole: Abilify (aripiprazole): Patients randomly assigned to aripiprazole received medication in pill form with dosing at 2mg, 5mg, 7mg, 10mg, 12mg or 15mg depending on their response.
- Placebo: placebo: Patients randomly assigned to placebo received pills/dosing made to look identical to the aripiprazole.
Period: Randomized Phase
Arm/Group | Aripiprazole | Placebo
Started | 31 | 31
Received More Than One Dose | 30 | 29
Completed | 15 | 6
Not Completed | 16 | 25
Not completed — Lack of Efficacy | 8 | 18
Not completed — Study nonadherence | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Participant reported having a rash | 1 | 0
Not completed — Emesis and enuresis | 0 | 1
Not completed — Oral/nasal twitching | 0 | 1
Period: Open Label Extension (OLE)
Arm/Group | Aripiprazole | Placebo
Started | 22 (Participants from aripiprazole group started OLE (eligible even if randomized period not completed).) | 21 (Participants from placebo group started OLE (eligible even if randomized period not completed).)
Completed | 17 | 15
Not Completed | 5 | 6
Not completed — Weight Gain | 1 | 0
Not completed — Drowsiness; Jittery | 0 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abilify Randomized Phase: Abilify (aripiprazole) : Patients randomly assigned to aripiprazole received medication in pill form with dosing at 2mg, 5mg, 7mg, 10mg, 12mg or 15mg depending on their response.
- Placebo Randomized Phase: Placebo: Patients randomly assigned to placebo received pills/dosing made to look identical to the aripiprazole.
- Total: Total of all reporting groups
Arm/Group | Abilify Randomized Phase | Placebo Randomized Phase | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 29 | 59
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 20 | 15 | 35
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: The Young Mania Rating Scale (YMRS) has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. Additional information is based upon clinical observations made during the course of the clinical interview. The items are selected based upon published descriptions of the core symptoms of mania. Each item o the YMRS is given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. There are well described anchor points for each grade of severity. Total score ranges from 0 to 60, with higher being more severe mania.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Abilify Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 30 | 29
Scores on a scale | 24.8 (6.8) | 21.6 (6.1)

2. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Abilify Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 30 | 29
Scores on a scale | 9.7 (9.2) | 16.2 (8.5)

3. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 1
Time Frame: Open-Label Extension - 6 weeks
Population: 22 patients in the Open-Label Extension (from initial Abilify) group and 21 patients in the Open-Label Extension (from initial placebo) group completed at least 1 week of the open-label extension (see participant flow). Due to missing data, data on 20 of those 22 and 18 of those 21 completed the YMRS and were available and included the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Open-Label Extension (Abilify): Participants entered the open-label extension phase of the study. They were originally assigned to the Abilify (aripiprazole) group in the 12-week randomized phase of the study.
  All participants in the open-label extension were taking Abilify (aripiprazole).
- Open-Label Extension (Placebo): Participants entered the open-label extension phase of the study. They were originally assigned to the placebo group in the 12-week randomized phase of the study.
  All participants in the open-label extension were taking Abilify (aripiprazole).
Arm/Group | Open-Label Extension (Abilify) | Open-Label Extension (Placebo)
Number analyzed (Participants) | 20 | 18
Scores on a scale | 5.73 (5.98) | 7.57 (5.12)

4. Secondary Outcome: Children's Depression Rating Scale-Revised (CDRS-R )
Description: The CDRS-R is a rating scale used to assess severity of depression and change in depressive symptoms in children and adolescents. The CDRS-R is a 17-item scale administered by clinician's in interviews with a child/parent(s). Each item is scored on a range of 1-5 or 1-7 with a total possible score of 17-113. A score greater or equal to 40 is indicative of depression and a score less than or equal to 28 is typically means few or no depressive symptoms.
Time Frame: Baseline
Population: There were 30 patients in the Abilify group and 29 patients in the placebo group who completed at least 1 week of the study as per the participant flow. As a result of missing data, data on 28 of 30 in the Abilify group and 28 of 29 in the placebo group were available and included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Aripiprazole Randomized Phase: Abilify (aripiprazole) : Patients randomly assigned to aripiprazole received medication in pill form with dosing at 2mg, 5mg, 7mg, 10mg, 12mg or 15mg depending on their response.
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
Scores on a scale | 33.7 (11.2) | 30.3 (10.4)

5. Secondary Outcome: CDRS-R Children's Depression Rating Scale-Revised
Description: as for outcome 4
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
Scores on a scale | 24.4 (7.5) | 25.9 (8.5)

6. Secondary Outcome: CDRS-R Children's Depression Rating Scale-Revised
Description: as for outcome 4
Time Frame: Open-Label Extension - 6 weeks
Population: 22 patients in the Open-Label Extension (from initial Abilify) group and 21 patients in the Open-Label Extension (from initial placebo) group completed at least 1 week of the open-label extension (see participant flow). Due to missing data, data on 20 of those 22 and 18 of those 21 completed the CDRS-R and were available and included the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Open-Label Extension (Abilify) | Open-Label Extension (Placebo)
Number analyzed (Participants) | 20 | 18
Scores on a scale | 21.5 (5.48) | 21.7 (5.54)

7. Secondary Outcome: Children's Global Assessment Scale (CGAS)
Description: Children's Global Assessment Scale (CGAS) is a scale that clinicians use in order to rate the general emotional and behavioral functioning of children and adolescents under age 18. The scoring range is either 1 to 100. Youth with higher scores indicate better functioning with 91-100 "Doing very well" to 1-10 Extremely impaired.
  The score should be calculated separate from diagnosis, treatment or prognosis.
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
Scores on a scale | 56.1 (6.7) | 57.5 (4.6)

8. Secondary Outcome: Children's Global Assessment Scale (CGAS)
Description: as for outcome 7
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
Scores on a scale | 67.1 (11.2) | 61.4 (8.7)

9. Secondary Outcome: Children's Global Assessment Scale (CGAS)
Description: as for outcome 7
Time Frame: Open-Label Extension - 6 weeks
Population: 22 patients in the Open-Label Extension (from initial Abilify) group and 21 patients in the Open-Label Extension (from initial placebo) group completed at least 1 week of the open-label extension (see participant flow). Due to missing data, data on 19 of those 22 and 18 of those 21 completed the CGAS and were available and included the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Open-Label Extension (Abilify) | Open-Label Extension (Placebo)
Number analyzed (Participants) | 19 | 18
Scores on a scale | 71.47 (8.49) | 69.72 (6.47)

10. Secondary Outcome: Clinical Global Impressions Scale (CGI-Severity)
Description: Clinical Global Impressions Scale (CGI-Severity) is a physician-administered assessment designed to track progress over time on a wide range of psychiatric disorders. The CGI-Severity or CGI-S consists of one question about the extent of a patient's mental illness at the time of the assessment. Using a 7-point rating scale, clinicians rate the severity of mental illness based on an average of observed and reported symptoms, behavior and function during the past 7 days. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
units on a scale | 4.2 (0.9) | 3.8 (0.8)

11. Secondary Outcome: Clinical Global Impressions Scale (CGI-Severity)
Description: as for outcome 10
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
units on a scale | 2.3 (1.4) | 3.0 (1.1)

12. Secondary Outcome: Clinical Global Impressions Scale (CGI-Severity)
Description: as for outcome 10
Time Frame: Open-Label Extension - 6 weeks
Population: 22 patients in the Open-Label Extension (from initial Abilify) group and 21 patients in the Open-Label Extension (from initial placebo) group completed at least 1 week of the open-label extension (see participant flow). Due to missing data, data on 20 of those 22 and 18 of those 21 completed the CGI-S and were available and included the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Open-Label Extension (Abilify) | Open-Label Extension (Placebo)
Number analyzed (Participants) | 20 | 18
Scores on a scale | 1.85 (.875) | 1.89 (.758)

13. Secondary Outcome: Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale IV or (ARS-IV)
Description: The Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale IV or (ARS-IV) is a clinician-scored rating scale used to track the frequency of ADHD symptoms during the previous 1-week period. The ARS-IV contains 18 questions--(9 focused on inattention, and 9 on hyperactivity-impulsivity.) Questions are answered in a way that best describes ADHD symptom frequency--Never or Rarely=0, Sometimes=1, Often=2, or Very Often=3. The clinician adds up the responses for a total score. Higher total scores indicate a greater degree of symptoms being present. As a result, the minimum score is 0, and the maximum score is 54.
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
units on a scale | 32.4 (12.4) | 36.8 (12.5)

14. Secondary Outcome: Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale IV or (ARS-IV)
Description: as for outcome 13
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aripiprazole Randomized Phase: Abilify (aripiprazole): Patients randomly assigned to aripiprazole received medication in pill form with dosing at 2mg, 5mg, 7mg, 10mg, 12mg or 15mg depending on their response.
Arm/Group | Aripiprazole Randomized Phase | Placebo Randomized Phase
Number analyzed (Participants) | 28 | 28
units on a scale | 21.0 (14.5) | 32.1 (14.3)

15. Secondary Outcome: Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale IV or (ARS-IV)
Description: as for outcome 13
Time Frame: Open-Label Extension - 6 weeks
Population: 22 patients in the Open-Label Extension (from initial Abilify) group and 21 patients in the Open-Label Extension (from initial placebo) group completed at least 1 week of the open-label extension (see participant flow). Due to missing data, data on 20 of those 22 and 17 of those 21 completed the ARS-IV and were available and included the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Open-Label Extension (Abilify) | Open-Label Extension (Placebo)
Number analyzed (Participants) | 20 | 17
Scores on a scale | 18.1 (14.0) | 28.1 (12.8)

ADVERSE EVENTS:
Groups:
- Abilify Randomized Phase: Abilify (aripiprazole): Patients randomly assigned to aripiprazole received medication in pill form with dosing at 2mg, 5mg, 7mg, 10mg, 12mg or 15mg depending on their response.
- Open Label Extension (Abilify): Previously randomized to Abilify group.
- Open Label Extension (Placebo): Previously randomized to placebo group.
Arm/Group | Abilify Randomized Phase | Placebo Randomized Phase | Open Label Extension (Abilify) | Open Label Extension (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 24/31 | 13/31 | 10/22 | 13/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abilify Randomized Phase (N=31) | Placebo Randomized Phase (N=31) | Open Label Extension (Abilify) (N=22) | Open Label Extension (Placebo) (N=21)
Headache (Nervous system disorders) | 15 | 12 | 8 | 5 — One case in the abilify group had a dosing reduction
Stomach ache (Gastrointestinal disorders) | 11 | 7 | 3 | 6 — One case in the abilify group had a dosing reduction
Sedation (General disorders) | 7 | 2 | 1 | 4 — One case in the placebo group had a dosing reduction
Increased appetite (General disorders) | 7 | 1 | 8 | 1 — Per study protocol as previously outlined
Emesis (Gastrointestinal disorders) | 7 | 0 | 6 | 1
Nausea (Gastrointestinal disorders) | 5 | 2 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 1 | 0
Fever (General disorders) | 4 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4 | 1 — Knee Pain, back ache
Dizziness (General disorders) | 4 | 2 | 0 | 1
Nasal Congestion (General disorders) | 3 | 1 | 1 | 0
Coughing (General disorders) | 4 | 0 | 2 | 0
Sore Throat (General disorders) | 2 | 1 | 1 | 0
Cold Symptoms (General disorders) | 2 | 1 | 3 | 0 — Runny nose, Sneezing
Weight Gain (General disorders) | 0 | 0 | 3 | 2
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 — Sinus infection
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Injury (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 2 — Broken leg, broken nose, heel injury
Athletes Foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Drowsiness (General disorders) | 0 | 0 | 0 | 11 — Tired, Tiredness, Fatigue, Going to bed early
Allergies (General disorders) | 0 | 0 | 0 | 5 — including nickel allergy
Feeling Cold (General disorders) | 0 | 0 | 0 | 3
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nose bleed (General disorders) | 0 | 0 | 0 | 2
Increased heart rate (Cardiac disorders) | 0 | 0 | 0 | 1
Decreased appetite (General disorders) | 0 | 0 | 0 | 1
Restlessness (General disorders) | 0 | 0 | 0 | 1
Influenza (General disorders) | 0 | 0 | 0 | 1 — Flu
Other (General disorders) | 0 | 0 | 0 | 1 — Can't remember music

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes